CLINICAL TRIAL: NCT02218541
Title: Fabrication of a Definitive Cad/Cam Titanium Abutment Prior to Guided Surgery: a Pilot Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-2376
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-05

CONDITIONS: Single Edentulous Space

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- abutment margin 0.5 mm subgingival (Other): when fabricating an abutment to support the crown, the margin will be placed 0.5 mm below the gumline
  Interventions: Device: abutment margin 0.5 mm subgingival
- abutment margin 1.5 mm subgingival (Other): when fabricating the abutment to support the crown, the margin will be placed 1.5 mm below the gumline
  Interventions: Device: abutment margin 1.5 mm subgingival

INTERVENTIONS:
Device: abutment margin 0.5 mm subgingival
  Arms: abutment margin 0.5 mm subgingival
Device: abutment margin 1.5 mm subgingival
  Arms: abutment margin 1.5 mm subgingival

SUMMARY:
The study will involve placing a dental implant through a guided surgery protocol developed using 3D CT technology. Because the implant position is planned digitally using the CT data from the patient, this allows investigation of an abutment that supports the implant crown and soft tissues to be fabricated prior to implant placement. In doing so, this makes the protocol for patient care simpler and faster. In fabricating the the abutment prior to surgery, the investigators will design the abutments at different heights below the gumline to see an optimal margin height for fabrication of the abutment prior to surgery. The study hypothesis is that more often the abutment margin placed just slightly below (.5mm) the gumline will be visible about half of the time while the abutment margin placed further under the gumline (1.5mm) will be visible only about 10% of the time. The optimal outcome is that at delivery and follow-up, the abutment margin will not show intraorally.

ELIGIBILITY:
Inclusion Criteria:

* partially edentulous with single edentulous space
* edentulous site where previous tooth has been extracted for at least two months
* minimum of 20 teeth present
* able to tolerate dental implant surgical and restorative procedures
* consent to participate in clinical trial

Exclusion Criteria:

* asa class 3+
* present drug use
* is pregnant or plans to become pregnant
* patients in need of lateral window sinus graft
* patients in need of grafting prior to implant placement
* patients in need of extensive grafting at time of implant placement
* tooth is present or extracted within the last 2 months
* history of IV bisphosphonate use or oral bisphosphonate use contraindicating dental implant therapy
* untreated caries or periodontal disease
* severe bruxism
* smoker within past 6 months
* unlikely to be able to comply with study procedures according to investigators
* known allergy to any materials used in dental implant surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg De Kok, DDS, Principal Investigator — University of North Carolina School of Dentistry
Locations (1):
- Graduate Prosthodontic Clinic, Dept. of Prosthodontics, UNC School of Dentistry, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Abutment Margin 0.5 mm Subgingival: When fabricating an abutment to support the crown, the margin will be placed 0.5 mm below the gumline abutment margin 0.5 mm subgingival
- Abutment Margin 1.5 mm Subgingival: When fabricating the abutment to support the crown, the margin will be placed 1.5 mm below the gumline abutment margin 1.5 mm subgingival
Period: Overall Study
Arm/Group | Abutment Margin 0.5 mm Subgingival | Abutment Margin 1.5 mm Subgingival
Started | 11 | 11
Completed | 5 | 9
Not Completed | 6 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Implant Failure | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abutment Margin 0.5 mm Subgingival | Abutment Margin 1.5 mm Subgingival | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 16
  >=65 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 7 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Abutment Margin Exposure > 0
Description: Margin exposure of the abutment between groups at 6 months post surgery.
Time Frame: up to 6 months post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Abutment Margin 0.5 mm Subgingival | Abutment Margin 1.5 mm Subgingival
Number analyzed (Participants) | 5 | 9
Participants | 0 | 0
Statistical Analysis 1: Comparison: Abutment Margin 0.5 mm Subgingival vs Abutment Margin 1.5 mm Subgingival; Test type: Other; p = 1.00, Fisher Exact — threshold for significance will be p-value <0.05

2. Secondary Outcome: Number of Participants With a Soft Tissue Response of Bleeding
Description: To assess the condition of the peri-implant mucosa, those with a soft tissue response of bleeding upon probing were counted. Fisher's exact test will be used after the site has been evaluated for presence of bleeding or not.
Time Frame: 6 months post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Abutment Margin 0.5 mm Subgingival | Abutment Margin 1.5 mm Subgingival
Number analyzed (Participants) | 5 | 9
Participants
  Yes bleeding | 3 | 8
  No bleeding | 2 | 1
Statistical Analysis 1: Comparison: Abutment Margin 0.5 mm Subgingival vs Abutment Margin 1.5 mm Subgingival; Test type: Other; p = 0.039, Binomial — This statistical analysis applies to Yes bleeding; The statistical analysis was changed during the analysis phase but the protocol was not amended to reflect this change

3. Secondary Outcome: Number of Participants With Provisional Crown Fit at Delivery
Description: To assess if the Provisional Crown was able to be cemented at time of abutment connection was reported as 'Yes' or 'No.'
Time Frame: 8 weeks post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Abutment Margin 0.5 mm Subgingival | Abutment Margin 1.5 mm Subgingival
Number analyzed (Participants) | 5 | 9
Participants
  Yes | 3 | 5
  No | 2 | 4
Statistical Analysis 1: Comparison: Abutment Margin 0.5 mm Subgingival vs Abutment Margin 1.5 mm Subgingival; Test type: Equivalence — No power calculation was done as this was a pilot study; p = 1.0, Binomial — This statistical analysis applies to Yes Provisional Crown fit; The statistical analysis was changed during the analysis phase but the protocol was not amended to reflect this change

ADVERSE EVENTS:
Time Frame: From the date of consent until six months after surgery
Groups:
- Abutment Margin 0.5 mm Subgingival: When fabricating an abutment to support the crown, the margin will be placed 0.5mm below the gumline abutment margin 0.5 mm subgingival
Arm/Group | Abutment Margin 0.5 mm Subgingival | Abutment Margin 1.5 mm Subgingival
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT02218541/Prot_SAP_000.pdf